CLINICAL TRIAL: NCT06048146
Title: A Prospective, Multicenter Randomized Controlled Study of the Application of Preoperative FOLFOXIRI Chemotherapy Combined With Lateral Lymph Node Dissection in Low- and Medium-lying Rectal Cancer With Lateral Lymph Node Metastasis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC2022L01
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Lymph Node Metastasis; Cancer of Rectum and Anus; Oxaliplatin; Intestinal Neoplasms; Gastrointestinal Neoplasms; Rectal Diseases; Rectal Neoplasms
MeSH Terms: conditions — Lymphatic Metastasis; Rectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Rectal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOXIRI and Lateral lymph node dissection (Experimental): Participants will
  * receive three cycles of chemotherapy with FOLFOXIRI regimen, and the specific dose was: irinotecan 150mg/m2, d1, Oxaliplatin 85mg/m2, d1, 5-Fu, 2400mg/m2, continuously pumped for 46 hours, repeated for 14 days.
  * After 3 cycles of chemotherapy, rectal MRI reexamination was performed, and the efficacy was evaluated using the RECIST method.
  * For cCR or cPR, another 2 cycles of chemotherapy will be performed, and CT and rectal MRI evaluations will be performed again after treatment. Radical rectal cancer surgery and LLND were performed 4-6 weeks after the last administration (unilateral or bilateral LLND was determined based on the metastasis of LLN before treatment).
  Interventions: Drug: Experimental: FOLFOXIRI and Lateral lymph node dissection; Drug: Preoperative long-term concurrent chemoradiotherapy and Lateral lymph node dissection
- Preoperative long-term concurrent chemoradiotherapy and Lateral lymph node dissection (Active Comparator): All patients received preoperative long-term concurrent chemoradiotherapy: radiotherapy for five weeks, five days a week (pelvic 2 Gy/ time, GT50 Gy), during which capecitabine (1650mg/m2/ day, orally divided twice). Intensity modulated radiotherapy was used. CT and rectal MRI were evaluated again 8-12 weeks after radiotherapy, followed by radical resection of rectal cancer plus LLND (unilateral or bilateral LLND was performed according to LLN metastasis before treatment).
  Interventions: Drug: Experimental: FOLFOXIRI and Lateral lymph node dissection; Drug: Preoperative long-term concurrent chemoradiotherapy and Lateral lymph node dissection

INTERVENTIONS:
Drug: Experimental: FOLFOXIRI and Lateral lymph node dissection — Irinotecan 150mg /m2, d1, oxaliplatin 85mg/m2, d1, 5-Fu, 2400mg/m2, pumped continuously for 46 hours and repeated for 14 days
Drug: Preoperative long-term concurrent chemoradiotherapy and Lateral lymph node dissection — Radiotherapy was administered five days a week (pelvic 2 Gy/ time, GT50 Gy) for five weeks with capecitabine (1650mg/m2/ day, orally divided into two doses). Intensity modulated radiotherapy (IMRT) was used

SUMMARY:
The goal of this clinical trial is to compare in newly diagnosed patients with resectable rectal cancer with lateral lymph node metastasis. This study aims to

* further verify the safety and efficacy of FOLFOXIRI three-drug regimen
* Using multiple omics techniques to identify and confirm specific molecular markers Participants will be treated with FOLFOXIRI three-drug combination regimen. Researchers will compare another group treated with conventional preoperative chemoradiotherapy to see if the experimental group is superior to the control group in terms of 3-year disease free survival, local recurrence rate, lateral lymph node positivity rate, and 5-year overall survival rate.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare in newly diagnosed patients with resectable rectal cancer with lateral lymph node metastasis. The main questions it aims to answer are:

* Evaluate the effectiveness and safety of Forfoxiri combined with lateral lymph node dissection, and optimize the treatment plan for rectal cancer patients with resectable lateral lymph node metastasis.
* Using multiple omics techniques to identify and confirm specific molecular markers for chemotherapy response, lateral lymph node metastasis, and distant metastasis in rectal cancer, in order to achieve the goal of precise treatment of lateral lymph node metastasis Participants will
* receive three cycles of chemotherapy with FOLFOXIRI regimen, and the specific dose was: irinotecan 150mg/m2, d1, Oxaliplatin 85mg/m2, d1, 5-Fu, 2400mg/m2, continuously pumped for 46 hours, repeated for 14 days.
* After 3 cycles of chemotherapy, rectal MRI reexamination was performed, and the efficacy was evaluated using the RECIST method.
* For cCR or cPR, another 2 cycles of chemotherapy will be performed, and CT and rectal MRI evaluations will be performed again after treatment. Radical rectal cancer surgery and LLND were performed 4-6 weeks after the last administration (unilateral or bilateral LLND was determined based on the metastasis of LLN before treatment).
* RECIST evaluates patients with SD, and if MRI evaluates rectal cancer patients without rectal fascia involvement (MRF -), they will undergo two cycles of triple drug combination chemotherapy. After treatment, CT and rectal MRI evaluations will be performed again. Rectal cancer radical surgery+LLND will be performed 4-6 weeks after the last administration.
* If MRF+is unable to complete R0 resection or RECIST evaluation of PD patients, in order to ensure the treatment effect of the patients, preoperative long-term synchronous radiotherapy and chemotherapy should be performed. Preoperative concurrent chemoradiotherapy regimen: Capecitabine (1650mg/m2/day, twice orally); Radiotherapy (pelvic cavity 2 Gy/dose, GT50 Gy); Intensity modulated radiation therapy is used for radiotherapy. CT and rectal MRI evaluations are performed again 8-12 weeks after radiotherapy, followed by rectal cancer radical surgery and LLND. If distant metastasis occurs during treatment, a second-line chemotherapy regimen can be chosen.

Researchers will compare another group (Capecitabine (1650mg/m2/day, oral administration twice) was used for long-term concurrent chemoradiotherapy before operation in all patients; Radiotherapy (pelvic cavity 2 Gy/dose, GT50 Gy). Intensity modulated radiation therapy is used for radiotherapy. CT and rectal MRI evaluation are performed again 8-12 weeks after radiotherapy, followed by rectal cancer radical surgery+LLND (unilateral or bilateral LLND is determined based on the LLN metastasis before treatment)) to see if the experimental group is superior to the control group in terms of 3-year disease free survival, local recurrence rate, lateral lymph node positivity rate, and 5-year overall survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old, gender is not limited;
* The clinical stage based on magnetic resonance imaging (MRI) is cT1-4aN+M0 (according to AJCC Cancer Staging Manual, 8th Edition, 2018).
* Meet the criteria for lateral lymph node metastasis (lymph node short diameter ≥7mm, or lymph node short diameter ≥5cm with uneven internal signals and no chemical shift effect, or irregular boundaries);
* The primary tumor was located in the rectum (hard tube proctoscopy indicated that the lower margin of the lesion was less than 10cm from the anus);
* Kastler score ≥70, ECOG score 0 or 1;
* Meet the following laboratory diagnostic indicators: hemoglobin ≥100g/L, white blood cells ≥3.5×109

  /L, neutrophil ≥1.5×109/L, platelet ≥100×109/L; Creatinine ≤1.5× upper limit of normal (UNL); Urea nitrogen (BUN) ≤1.5 upper limit of normal (UNL) alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤2.5×UNL, alkaline phosphatase (ALP) ≤2.5×UNL, total bilirubin (Tbil) ≤2.5×UNL; Urinary protein (-); Clotting time is normal.
* Patients with primary locally advanced rectal cancer required that they had not received surgery, radiotherapy, chemotherapy or other antitumor therapy from diagnosis to enrollment; No previous pelvic radiation;
* Subjects voluntarily join the study and sign the informed consent.

Exclusion Criteria:

* A history of malignancy at other sites, excluding curable non-melanic skin cancer and carcinoma in situ of the cervix;
* Unable to complete MRI;
* Preoperative examination indicated the need for combined organ resection;
* Allergic to 5-Fu and platinum drugs; Inability to swallow oral medications;
* The patient is under thrombolytic or anticoagulant therapy, has bleeding diathesis or coagulation dysfunction, or has occurred in the past year Aneurysm, stroke, transient ischemic attack, arteriovenous malformation;
* After renal history, urine test found proteinuria or clinical renal function was obviously abnormal;
* History of digestive tract fistula, perforation or severe ulcer;
* Active infection is present; Clinically significant cardiac disease (e.g., uncontrolled hypertension (160/110) mm Hg blood pressure, any history of myocardial infarction, unstable angina), NYHA class Ⅱ congestive heart failure, unstable symptomatic arrhythmias, or class II peripheral vascular disease. Myocardial infarction and cerebrovascular accident occurred within 6 months before enrollment;
* Participating in other clinical trials currently or within 4 weeks prior to enrollment;
* long-term adverse drug history, drug addiction history of mental disorders;
* Other cases where the examiner considers from the registration study that there are good reasons for non-conformity: if there are potential inconsistencies with the clinical protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
3 year disease free survival | From after surgery to three years after surgery
  The time between the initiation of a treatment and the recurrence of the disease or death (from any cause)

CONTACTS AND LOCATIONS:
Overall Officials: jianwei liang, M.D., Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing, Beijing Municipality, China